CLINICAL TRIAL: NCT05227222
Title: Evaluation of Positive Expiratory Pressure Device (PEP-device) for Treatment of Swimming Induced Pulmonary Edema (SIPE) - a Randomized Single-blinded Controlled Study
Brief Title: PEP-device for Treatment of Swimming-induced Pulmonary Edema (SIPE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hårdstedt, Dr. Maria Hårdstedt, PhD, Specialist Internal Medicine, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIPE PEP-device001
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Swimming Induced Pulmonary Edema (SIPE); Pulmonary Edema; Lung Diseases
Keywords: positive expiratory pressure; therapeutics; ultrasonography; oximetry
MeSH Terms: conditions — Pulmonary Edema; Lung Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEP-device (Experimental): Positive expiratory pressure device: continuous treatment with PEP-device breathing air for 20 minutes followed by 10 minutes rest and assessment. Inspiration through nose/mouth, expiration through device.
  Interventions: Device: PEP-device
- spontaneous recovery (No Intervention): Control group: Resting and breathing air for 20 + 10 minutes.

INTERVENTIONS:
Device: PEP-device — PEP-device
  Arms: PEP-device

SUMMARY:
In swimming induced pulmonary edema (SIPE), there is a lack of knowledge regarding optimal treatment. The present study was designed to assess the benefit of treatment with positive expiratory pressure device (PEP-device) compared to spontaneous recovery in patients with SIPE without hypoxia in the out-of-hospital environment.

DETAILED DESCRIPTION:
Swimming induced pulmonary edema (SIPE) is an unusual condition affecting otherwise healthy swimmers. SIPE is characterized by acute onset of dyspnea and cough, excessive sputum and occasionally hemoptysis when swimming in open water. The condition usually resolves spontaneously within 48 hours, but may result in serious illness and require emergency care. Case reports describe acute treatment with or without oxygen in combination with diuretics, beta-agonist-inhalation or continuous positive airway pressure (CPAP). Evidence for optimal treatment strategy is lacking. Oxygen treatment might not be appropriate for patients with SIPE presenting without hypoxia. It is unknown if positive airway pressure accelerates recovery in SIPE.

This study intends to determine whether treatment with positive expiratory pressure (PEP) applied by PEP-device accelerates increase of oxygen saturation compared to spontaneous recovery in patients presenting with SIPE without hypoxia. The aim is to treat patients on site without involving hospital care. We study a large cohort of approximately 12 000 swimmers during Vansbrosimningen, Sweden's biggest annual open water event with a yearly incidence of SIPE about 0,4%.

Adult patients clinically diagnosed with SIPE and oxygen saturation ≥92% are randomly assigned to 2 groups: (1) PEP-device for 20 minutes or (2) control group with spontaneous recovery without active treatment for 20 minutes. Assessment with outcome measures is taken 10 minutes after intervention/control. Primary endpoint: oxygen saturation (%) by pulse oxymetry.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of swimming induced pulmonary edema (SIPE) with need of acute treatment
* peripheral oxygen saturation ≥92%
* 18 years or older
* informed consent

Exclusion Criteria:

* declined consent
* suspected acute coronary syndrome
* severe asthma diagnosed together with pulmonary edema with requirement of beta-agonist-inhalation prior to treatment of pulmonary edema
* hemodynamic instability or decreased consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Absolute peripheral oxygen saturation (%) after treatment | after 20 min treatment followed by 10 min rest
  Peripheral oxygen saturation % (continuous variable) measured by peripheral pulse oximetry

SECONDARY OUTCOMES:
Change in absolute peripheral oxygen saturation (%) before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Change in peripheral oxygen saturation % (continuous variable) measured by pulse oximetry before and after treatment
Recovery (yes/no) after treatment | after 20 min treatment followed by 10 min rest
  Recovery, defined by "peripheral oxygen saturation >95% after treatment" or no recovery, defined by "peripheral oxygen saturation ≤95% after treatment"
Interstitial syndrome assessed by lung ultrasound (yes/no) after treatment | after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Bilateral or unilateral presence of two or more positive regions define positive interstitial syndrome
Absolute number of regions presenting B-lines on lung ultrasound after treatment | after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions.
Change in absolute number of regions presenting B-lines on lung ultrasound before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions. Change in absolute number of regions presenting B-lines on lung ultrasound before and after treatment
Change in patient reported outcome measures before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Six different patient reported outcome measures assessed by numerical rating scale (NRS; min-max 0-10): cough, sputum, air hunger, breathing effort, tightness in chest, anxiousness. The patients will assess symptoms prior to and after treatment
Admission to hospital (yes/no) | 1 hour
  Admission to hospital within or after a maximal treatment time of 1 hour
Total treatment time | 1 hour
  Total treatment time until oxygen saturation ≥96% is reached

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Clinical Research Dalarna, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No